CLINICAL TRIAL: NCT06837753
Title: Does Hamstring Stretching Effective on Nonspecific Low Back Pain?"
Brief Title: Hamstring Stretching Effective on Nonspecific Low Back Pain
Acronym: Hams
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Eylül Pınar KISA, Investigators, Biruni University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hamstring
Record Dates: First submitted 2023-12-13; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- exercise group (Experimental): Exercise program and 3 way hamstring strech will be applied.
  Interventions: Other: Exercise
- control group (Other): Just Exercise program will be applied.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — It consist of traditional exercises.

SUMMARY:
Low back pain is one of the most common complaints in the world and can be considered a universal health problem for humanity. Low back pain is a multifactorial disease with multiple etiologies. Risk factors are difficult to identify. It is reported in the literature that 70-80% of the world's population has low back pain at some point in their lives, and 95% of this pain is mechanical. Mechanical low back pain (MBA) can be described as a clinical picture that develops as a result of overuse, strain, traumatization or deformation of the structures that make up the spine. In order to define low back pain mechanically, all organic causes such as inflammatory, infectious, tumoral, metabolic causes, fractures and pain reflected from internal organs must be excluded. The most common diseases that cause low back pain are; They are caused by mechanical factors and degenerative diseases. Mechanical and static stresses can lead to joint blockage, restricting the range of motion of the joint along with pain. Non-Specific many factors affect low back pain. Kim and Shin reported that asymmetry of hip extension range of motion of both hip joints was associated with nonspecific low back pain rather than simple hip extension range of motion, and they found that limiting hip extension was compensatory.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complaints of low back pain,
* NLBP for at least 12 weeks,
* finger-to-ground distance greater than 0 cm; a passive straight-leg raising -(SLR) angle of less than 80°, measured with a hand-held goniometer;
* normal mobility of the hip;
* passive knee extension ≥25°,
* VAS score between 3 and 7 will be included.

Exclusion Criteria:

* People with a history of hamstring injury in the last two years,
* fractures in the spine or lower extremities,
* pregnancy,
* leg length difference of more than 2 cm,
* and obesity will be excluded from the study.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Pain status | 0-8 week
  Pain status Patients pain status were evaluated with VAS between 0 and 10 for low back pain during movement. (No pain at 0 points, severe pain at 10 points)
Flexibility assessment | 0-8 week
  During Single Leg Raise, subjects were asked to indicate (by pushing a button) the beginning of pain or an unpleasant tension sensation in the dorsal part of the thigh off the knee. This first sensation of pain was recorded as a function of the pelvic-femoral angle. Subjects were also instructed to push the button and to say "stop" when they could no longer tolerate more movement or stretch; at that point, the leg raise was stopped. The stretch tolerance was defined by the extensibility of the hamstrings. Note that the subjects stopped the leg raise.

SECONDARY OUTCOMES:
Functionality index | 0-8 week
  Functional Rating Index (FDI) was obtained by combining similar structures of the neck disability index and the Osweestry low back pain disability index, and its validity and reliability have been proven. The validity and reliability of the Turkish version of this survey was conducted by Bayar et al. in 2004. FDI consists of 10 parts that measure the function of the spinal musculoskeletal (waist, neck pain) system and pain. Eight address activities of daily living that may be affected by the spinal condition. Two of them address 2 different characteristics of pain. Using a 5-choice scale for each item, the amount of current pain or perceived ability to function is ranked by selecting 5 response points. 0=no pain or full function, 1=mild pain or mild limitation, 2=moderate pain or moderate limitation, 3=severe pain or severe limitation, 4=worst pain or inability to function. Scoring varies between 0-40, and as the score increases, functional status worsens
FUNCTIONAL STATUS | 0-8 week
  It consists of 10 questions, each scored between 0 and 5, assessing pain, personal care, lifting loads, walking, sitting, standing, sleeping, social life, traveling and the degree of change in pain. The maximum score is 50 and the total score is multiplied by two and the result is given as a percentage. Evaluation; It is done with the formula score/total score (50) x 100 = %. This form is a form with proven validity and reliability in Turkish for patients with chronic low back pain, used to evaluate treatment results and compare different treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Eylül Pınar Kısa, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No